CLINICAL TRIAL: NCT03234972
Title: A Randomized, Multicenter, Open-label, Phase 3 Study to Compare Daratumumab, Bortezomib, and Dexamethasone (DVd) vs Bortezomib and Dexamethasone (Vd) in Chinese Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study to Compare Daratumumab, Bortezomib, and Dexamethasone (DVd) vs Bortezomib and Dexamethasone (Vd) in Chinese Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104378; 54767414MMY3009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Daratumumab, Velcade, and Dexamethasone (DVd) (Experimental): Participants will receive daratumumab weekly for the first 3 cycles, every 3 weeks (q3w) on Day 1 of Cycles 4-9 as an intravenous (IV) infusion at a dose of 16 milligram per kilogram (mg/kg) or will have the option to switch to daratumumab subcutaneously (SC) on Day 1 of any cycle, and then every 4 weeks (q4w) thereafter, Velcade at a dose of 1.3 milligram per square meter (mg/m^2) subcutaneous (SC) on Days 1, 4, 8 and 11 of each 21-day cycle (up to 8 treatment cycles) and dexamethasone (Dex) orally (PO) at 20 milligram (mg) on Days 1, 2, 4, 5, 8, 9, 11 and 12 of the 8 Velcade treatment cycles.
  Interventions: Drug: Daratumumab; Drug: Velcade; Drug: Dexamethasone
- Arm B: Velcade and Dexamethasone (Vd) (Experimental): Participants will receive Velcade SC at a dose of 1.3 mg/m^2 SC on Days 1, 4, 8 and 11 of each 21-day cycle and Dex 20 mg PO on Days 1, 2, 4, 5, 8, 9, 11, 12 (up to 8 cycles). Participants who have sponsor-confirmed disease progression while being treated with Vd or on observation, will be offered the option for treatment with daratumumab monotherapy (16 mg/kg weekly for Cycles 1 and 2, every other week for Cycles 3 to 6, and every 4 weeks for Cycles 7 and onwards until disease progression, unacceptable toxicity, pregnancy, loss of follow-up, withdrawal of consent, or death [each cycle is 28 days]), if recommended by the site investigator.
  Interventions: Drug: Daratumumab; Drug: Velcade; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered on Day 1 of Cycles 4-9, and then q4w thereafter.
Drug: Velcade — Velcade will be administered at a dose of 1.3 mg/m^2 SC on Days 1, 4, 8 and 11 of each 21-day cycle.
Drug: Dexamethasone — Dex will be administered orally at 20 mg on Days 1, 2, 4, 5, 8, 9, 11 and 12 of the first 8 Velcade treatment cycles.

SUMMARY:
The primary purpose of this study is to compare the efficacy of daratumumab when combined with Velcade (bortezomib) and dexamethasone (DVd) to that of Velcade and dexamethasone (Vd), in terms of progression free survival (PFS) in Chinese participants with relapsed or refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma (MM) as defined by the criteria: monoclonal plasma cells in the bone marrow greater than or equal to (>=) 10 percent (%) at some point in the participant's disease course or presence of a biopsy-proven plasmacytoma
* Received at least 1 prior line of therapy for MM
* Documented evidence of progressive disease (PD) based on investigator's determination of response as defined by the International Myeloma Working Group (IMWG) criteria on or after their last regimen
* Achieved a response (partial response [PR] or better based on investigator's determination of response by the IMWG criteria) to at least 1 prior regimen
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2

Exclusion Criteria:

* Received daratumumab or other anti-CD38 therapies
* Refractory to Velcade, or another proteasome inhibitor (PI), like ixazomib and carfilzomib (ie, participant had progression of disease while receiving Velcade therapy or within 60 days of ending Velcade therapy, or another PI, like ixazomib and carfilzomib, etc)
* Intolerant to Velcade (that is [ie], discontinued due to any adverse event while on Velcade treatment)
* Planning to undergo a stem cell transplant prior to progression of disease on this study, that is ie, these participants should not be enrolled in order to reduce disease burden prior to transplant
* History of malignancy (other than MM) within 3 years before the date of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of randomization to either progressive disease (PD) or death, whichever occurs first (approximately up to 4.5 years)
  PFS is duration from date of randomization to either PD (as per international myeloma working group [IMWG] criteria) or death whichever occurs first. PD: Increase of 25 percent (%) from lowest response value in one of following: Serum M-component and urine M-component (absolute increase must be greater than or equal to [>=]0.5 gram per deciliter [g/dL] and >=200 mg/24 hours respectively); Only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be >10 mg/dL); only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell (PC) percentage (absolute percentage must be >=10%); definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11.5 mg/dL).

SECONDARY OUTCOMES:
Time to Disease Progression (TTP) | From the date of randomization to the date of first documented evidence of PD (approximately up to 4.5 years)
  TTP is defined as time from date of randomization to date of first documented evidence of PD. PD per IMWG criteria: Increase of 25 % from lowest response value in one of following: Serum M-component and urine M-component (absolute increase must be >=0.5 g/dL and >=200 mg/24 hours respectively); Only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase must be greater than [>]10 mg/dL); only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC percentage (absolute percentage must be >=10%); definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11.5 mg/dL).
Overall Response Rate (ORR) | Approximately up to 4.5 years
  ORR is percentage of participants who achieve partial response (PR) or better (stringent complete response [sCR], complete response [CR], VGPR), according to the IMWG criteria, during the study or during follow up. PR: >=50% reduction of serum M-protein, >=90% reduction in 24 hour urinary M-protein or to <200 mg/24 hours; if serum and urine M-protein are not measurable, >=50% decrease in difference between involved and uninvolved FLC levels; if serum and urine M-protein and serum free light assay is not measurable, >=50% reduction in bone marrow PC, with baseline bone marrow PC percentage >=30%; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; VGPR: serum and urine M-component detectable by immunofixation or >=90.0% reduction in serum M-protein and urine M-protein <100mg/24 hours; CR: negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5.0% PCs in bone marrow; sCR: CR plus normal FLC ratio and absence of clonal PCs.
Percentage of Participants With a Very Good Partial Response (VGPR) or Better | Approximately up to 4.5 years
  VGPR or better rate defined as the percentage of participants achieving VGPR and CR (including sCR) according to the IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or >=90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours; CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow; sCR: CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry.
Time to Response | From the date of randomization and the first efficacy evaluation that the participant has met all criteria for response (PR or better rate) (approximately up to 4.5 years)
  Time to response, defined as the time between the date of randomization and the first efficacy evaluation that the participant has met all criteria for response (PR or better rate). IMWG criteria for PR: >=50% reduction of serum M-protein, >=90% reduction in 24 hour urinary M-protein or to <200 mg/24 hours; if serum and urine M-protein are not measurable, >=50% decrease in difference between involved and uninvolved FLC levels; if serum and urine M-protein and serum free light assay is not measurable, >=50% reduction in bone marrow PC, with baseline bone marrow PC percentage >=30%; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; VGPR: serum and urine M-component detectable by immunofixation or >=90.0% reduction in serum M-protein and urine M-protein <100mg/24 hours; CR: negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5.0% PCs in bone marrow; sCR: CR plus normal FLC ratio and absence of clonal PCs.
Duration of Response | From the date of initial documentation of a response (PR or better rate) to the date of first documented evidence of PD (approximately up to 4.5 years)
  Duration of response will be calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of PD, as defined in the IMWG criteria. IMWG criteria for PR: >=50% reduction of serum M-protein and reduction in 24 hour urinary M-protein by >=90% or to <200 mg/24 hours, if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria,If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow PCs is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30% in addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Overall Survival | From date of randomization to the date of the participant's death (approximately up to 4.5 years)
  Overall survival is measured from the date of randomization to the date of the participant's death.
Change From Baseline in Euro Quality of Life 5-Dimensions 5-Level (EQ-5D-5L) Utility Score | Baseline up to Weeks 8 and 16 post PD (Approximately up to 4.5 years)
  EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 dimensions are used to compute a single utility score ranging from zero (0.0) to 1 (1.0), with higher values representing better general health status of the individual.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Baseline up to Weeks 8 and 16 post PD (Approximately up to 4.5 years)
  EORTC QLQ-C30 is a cancer-specific measure of health-related quality of life (HRQoL) that includes 30 items resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 Global Health Status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The recall period is 1 week (the past week). Scores are transformed to a 0 to 100 scale. A higher score for the global health status scale represents greater quality of life, a higher score for a functional scale represents greater functioning, and a higher score for a symptom scale/item represents more symptomatology/problems.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (27):
- China (25):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People s Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital Si Chuan University, Chengdu
  - Xinqiao Hospital of the Third Military Medical University, Chongqing
  - Fujian Meidical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Nanfang Hospital, Guangzhou
  - First Affiliated Hospital Medical School of Zhejiang University, Hangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Changzheng Hospital, Shanghai
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - First Affiliated Hospital SooChow University, Suzhou
  - Tianjin cancer hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - Tangdu Hospital, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

REFERENCES:
- [Derived] Fu W, Li W, Hu J, An G, Wang Y, Fu C, Chen L, Jin J, Cen X, Ge Z, Cai Z, Niu T, Qi M, Gai X, Li Q, Liu W, Liu W, Yang X, Chen X, Lu J. Daratumumab, Bortezomib, and Dexamethasone versus Bortezomib and Dexamethasone in Chinese Patients With Relapsed or Refractory Multiple Myeloma: Updated Analysis of LEPUS. Clin Lymphoma Myeloma Leuk. 2023 Jan;23(1):e51-e58. doi: 10.1016/j.clml.2022.10.007. Epub 2022 Oct 23. PMID 36402700
- [Derived] Lu J, Fu W, Li W, Hu J, An G, Wang Y, Fu C, Chen L, Jin J, Cen X, Ge Z, Cai Z, Niu T, Qi M, Sun S, Gai X, Liu W, Liu W, Yang X, Huang X. Daratumumab, Bortezomib, and Dexamethasone Versus Bortezomib and Dexamethasone in Chinese Patients with Relapsed or Refractory Multiple Myeloma: Phase 3 LEPUS (MMY3009) Study. Clin Lymphoma Myeloma Leuk. 2021 Sep;21(9):e699-e709. doi: 10.1016/j.clml.2021.04.012. Epub 2021 Apr 24. PMID 34108127